CLINICAL TRIAL: NCT02389582
Title: Effects of LMWH Versus Dabigatran on Platelet Aggregation in Patients With Stable Coronary Artery Disease
Brief Title: Effects of Low Molecular Weight Heparin Versus Dabigatran on Platelet Aggregation in Patients With Stable Coronary Artery Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SDC 3877/13/002
Record Dates: First submitted 2014-12-04; First posted 2015-03-17 (Estimated); Last update posted 2016-04-29 (Estimated); Status verified 2014-08

CONDITIONS: Coronary Disease
Keywords: platelet function; dabigatran;enoxaparin
MeSH Terms: conditions — Coronary Disease | interventions — Dabigatran; Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dabigatran (Experimental): Dabigatran 150mg twice a day for five days
  Interventions: Drug: Dabigatran
- Enoxaparin (Active Comparator): Enoxaparin 1mg/kg/day twice a day for five days
  Interventions: Drug: Enoxaparin

INTERVENTIONS:
Drug: Dabigatran — Use for 5 days
  Other Names: Pradaxa
  Arms: Dabigatran
Drug: Enoxaparin — Use for 5 days
  Other Names: Clexane
  Arms: Enoxaparin

SUMMARY:
Anticoagulation with heparin is indicated in several situations, such as acute coronary disease (in combination with antiplatelet therapy) for the prevention and treatment of venous thromboembolism and situations with high risk of thromboembolism. Recently, the latest trials on anticoagulation for stroke prevention on atrial fibrillation have shown an increased risk for acute mycardial infarction on patients submitted to new oral anticoagulants, such as dabigatran. The mechanism is still unclear, however, in this context, some previous studies about interaction between anticoagulants ( mainly heparin) and platelet aggregation have shown conflicting results: while some suggest an inhibitory effect of heparin on platelet function, others suggest that heparin could promote an increase in platelet activation. The present study aims to assess the effects of the LMWH Enoxaparin and direct thrombin inhibitor, Dabigatran, on platelet aggregation, studied and compared by different methods in patients with chronic coronary artery disease (CAD).

DETAILED DESCRIPTION:
This is a prospective and open study. We will include 29 patients with chronic CAD, stable, using ASA. All patients will receive the same medications in effective doses recommended at each stage of the study, so that every individual is his self-control, the Enoxaparin will be administrated at a dose of 1mg/kg twice a day and Dabigatran at a dose of 150mg twice a day. Study Design: Phase 1 : There will be a first collection of blood samples from all patients at baseline for laboratory tests, then the patient will receive Dabigatran for 5 days and laboratory tests including platelet aggregation will be made, among others. After a 30 days washout period, enoxaparin will be administrated for 5 days and in the 6st day, the same laboratory tests, including platelet aggregation, will be performed.

ELIGIBILITY:
Inclusion Criteria:

Age > 18 years old Coronary artery disease, defined as previous myocardial infarction and/or coronary angioplasty and/or Coronary Artery Bypass Graft (CABG) surgery and/or coronariography showing obstruction of at least 50 % in one of major epicardial vessels Treatment with Acetylsalicylic Acid (ASA) 100 mg/day

Exclusion Criteria:

Use in the last 7 days of oral anticoagulant or any other antiplatelet drug beside ASA Active bleeding Pregnancy or woman of childbearing age without contraceptive method Hemoglobin < 10 g/dL or hematocrit < 30 %, hematocrit > 50 %, platelets < 100.000/mm3 or > 500.000/mm3; creatinin clearance < 50 ml/minute Percutaneous coronary intervention (PCI) on the last 30 days before randomization (or PCI on the last year when drug-eluted stents are used); CABG surgery on the last 90 days; acute coronary syndrome on the last 60 days Active malignant neoplasm Active peptic ulcer disease on the last 60 days or upper gastrointestinal bleeding any time in life Refuse to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-05; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Platelet Aggregability | 5 days after starting the drug
  Comparing PLATELET AGGREGABILITY values through Multiplate test between patients on aspirin, assigned to the groups dabigatran and enoxaparin.

SECONDARY OUTCOMES:
Change from Baseline Platelet Aggregability with other aggregability test | 5 days after starting the drug
  Comparing PLATELET AGGREGABILITY values through Verify Now test (units=ARU) between patients on aspirin assigned to the groups dabigatran and enoxaparin

OTHER OUTCOMES:
Comparing the main outcome on pre-specified subgroups | 5 days after starting the drug
  elderly (age > 65 yrs-old) versus non-elderly male versus female smoking versus non-smoking patients diabetic versus non-diabetic
Correlate platelet aggregability and inflammation markers | 5 days after starting the drug

CONTACTS AND LOCATIONS:
Overall Officials: José C Nicolau, PhD, Principal Investigator — InCor Heart Institute - University of São Paulo
Locations (1):
- InCor Heart Institute, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Arantes FBB, Menezes FR, Franci A, Barbosa CJDG, Dalcoquio TF, Nakashima CAK, Baracioli LM, Furtado RHM, Nomelini QSS, Ramires JAF, Kalil Filho R, Nicolau JC. Influence of Direct Thrombin Inhibitor and Low Molecular Weight Heparin on Platelet Function in Patients with Coronary Artery Disease: A Prospective Interventional Trial. Adv Ther. 2020 Jan;37(1):420-430. doi: 10.1007/s12325-019-01153-8. Epub 2019 Nov 22. PMID 31758517